CLINICAL TRIAL: NCT01808495
Title: Function and Modulation of Fibulin-1 Assembly in Nucleus of Corneal Fibroblasts
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Tsan-Chi Chen, Department of Ophthalmology, Far Eastern Memorial Hospital
Other Study IDs: FEMH-IRB-101002-F; NSC101-2320-B-418-002 (Other Grant/Funding Number: NSC101-2320-B-418-002)
Record Dates: First submitted 2012-09-13; First posted 2013-03-11 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Function of Mitomycin C in Cornea
Keywords: Human corneal fibroblasts; Fibulin-1; Nuclear accumulation
MeSH Terms: interventions — Mitomycin

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Mitomycin C

SUMMARY:
The purpose of this study is to investigate the role of nuclear Fibulin-1 (FBLN1) in Human Corneal Fibroblasts under treatment of mitomycin C (MMC).

ELIGIBILITY:
Inclusion Criteria:

* The frozen storage cells in liquid nitrogen were amplified from the residual corneal rim of the donors with more than 20 years old following penetrating keratoplasty.

Exclusion Criteria:

* The donors were younger than 20 years old.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The original cell sources were collected from the donors with more than 20 years old following penetrating keratoplasty. After successfully amplified from the residual corneal rim following penetrating keratoplasty in the previous projects, human corneal fibroblasts (HCFs) were reserved in liquid nitrogen tank and were thawed for this study under in vitro cultivation and application.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-07 (Actual); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Modification of nuclear Fibulin-1 accumulation in suppressing gene expression | 3 days post mitomycin C treatment

CONTACTS AND LOCATIONS:
Overall Officials: Tsan-Chi Chen, PhD, Principal Investigator — Far Eastern Memorial Hospital